CLINICAL TRIAL: NCT06071702
Title: IonMAN II Trial- Early Feasibility Study of the IoNIR Ridaforolimus-Eluting Coronary Stent System
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated in any site. Sponsor decided not to start the study
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IoNIR-002
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Coronary Stenosis; Coronary Artery Disease
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- IoNIR Ridaforolimus-Eluting Coronary Stent (Experimental): IoNIR Ridaforolimus-Eluting Coronary Stent System
  Interventions: Device: IoNIR Ridaforolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: IoNIR Ridaforolimus-Eluting Coronary Stent System — The IoNIR Ridaforolimus-Eluting Coronary Stent System is a sterile single-use device/drug combination product, comprised of a cobalt chromium (CoCr) alloybased stent coated with a bioresorbable polymer mesh which is embedded with drug, mounted on a Rapid Exchange (RX) delivery system.

SUMMARY:
This is a prospective, multi-center, single-arm, open-label, early feasibility study to provide preliminary evidence for the safety and efficacy of the novel IoNIR stent system

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient with an indication for PCI including NSTEMI (biomarkers have peaked or are falling), angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80, Pd/Pa≤0.91or iFR, RFR, DFR, DPR≤0.89 must be present).
3. Non-target vessel PCIs are allowed if performed >30 days prior to index procedure.
4. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.
5. Staged procedures are allowed as long as the IoNIR stent is implanted in the last procedure and at least 30 days have elapsed between the previous procedure and the IoNIR PCI.
6. A maximum of two vessels and up to two lesions may be treated (two lesions separated by up to 10mm that can be covered by a single stent are considered as one lesion).
7. Lesions requiring scoring/cutting and/or rotational/orbital atherectomy and/or intra-vascular lithotripsy are allowed.
8. Overlapping stents are allowed.
9. Target lesion must be in a major native coronary artery with visually estimated diameter of ≥2.5 mm to ≤4.0 mm and lesion length of up to 40 mm, and appropriate size IoNIR stents are available.

Exclusion Criteria:

* 1. ST Segment Elevation MI within past 30 days. 2. NSTEMI with biomarkers that have not peaked. 3. Significant valvular disease or planned valvular intervention. 4. PCI within the 30 days preceding the baseline procedure. 5. PCI in the target vessel within 12 months of the baseline procedure. 6. Planned staged procedures (coronary or valvular), where the study stent is implanted in the first stage.

  7. Brachytherapy in conjunction with the baseline procedure. 8. Known history of stent thrombosis. 9. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.

  10. Subject is intubated. 11. Known LVEF <30%. 12. Contraindication to DAPT for 6 months in non-ACS patients and 12 months in ACS patients (including planned surgeries that cannot be delayed).

  13. Subject has an indication such as atrial fibrillation for oral anticoagulation/prolonged heparinization (i.e., use of coumadin/DOAC (NOAC) or prolonged enoxaparin/heparin therapy is not allowed).

  14. eGFR <60 mL/min. 15. Hemoglobin <10 g/dL. 16. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3. 17. White blood cell (WBC) count <3,000 cells/mm3. 18. Clinically significant liver disease. 19. Active peptic ulcer or active bleeding from any site. 20. Bleeding from any site within the previous 8 weeks requiring active medical or surgical attention.

  21. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.

  22. History of bleeding diathesis or coagulopathy and patients that refuse blood transfusions.

  23. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.

  24. Known allergy to the study stent components (cobalt, nickel, chromium, molybdenum, platinum, PDLG, PLC, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).

  25. Known allergy to protocol-required concomitant medications such as aspirin, or P2Y12 inhibitors (clopidogrel, prasugrel, and ticagrelor), heparin and bivalirudin, or iodinated contrast allergy that cannot be adequately pre-medicated.

  26. Any co-morbid condition that may cause non-compliance with the protocol (e.g., dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g., cancer, severe heart failure, severe lung disease).

  27. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.

  28. Women who are pregnant or breastfeeding. 29. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).

  30. Patient has received an organ transplant or is on a waiting list for an organ transplant.

  31. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.

  32. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

  33. Complex lesions including severely calcified lesions, presence of visible thrombus, chronic total occlusions, bifurcation lesions (side branch diameter ≥2.0 mm), tortuous lesions, restenotic lesions, left main lesions, ectasia, aneurysm and any bypass graft lesions.

  34. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure.

  35. Ostial lesions within 3 mm of origin of LAD, LCx, lesions in the LM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
In-stent Late Loss (LL) | 13 months
  In-stent Late Loss (LL) at 13 months assessed by quantitative coronary angiography (QCA) (Minimal Lumen Diameter (MLD) post-procedure - MLD follow-up (US patients only))
Target Lesion Failure | 1 year
  Target Lesion Failure (composite of cardiovascular death, target vessel-related myocardial infarction, or ischemia-driven target lesion revascularization)

SECONDARY OUTCOMES:
Major adverse cardiac events | 30 days, 6 months, 1,2,3,4,5 years
  Major adverse cardiac events (MACE; the composite rate of cardiovascular death, any MI or ischemia-driven target lesion revascularization (TLR)).
All-cause mortality | 30 days, 6 months, 1,2,3,4,5 years
  All-cause mortality
Cardiovascular death | 30 days, 6 months, 1,2,3,4,5 years
  Cardiovascular death
Myocardial infarction | 30 days, 6 months, 1,2,3,4,5 years
  Myocardial infarction
Target vessel related MI | 30 days, 6 months, 1,2,3,4,5 years
  Target vessel related MI
Target Lesion Failure | 6 months, 2, 3, 4, 5 years
  Target Lesion Failure
Ischemia-driven TLR | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Ischemia-driven TLR
Ischemia-driven Target Vessel Revascularization | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Ischemia-driven Target Vessel Revascularization
Stent thrombosis | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Stent thrombosis (ARC-2 definite and probable).
Acute Device Success | index procedure
  Acute Device Success (successful crossing and deployment with residual QCA DS <30%)
Luminal gain | 13 months - US patients only
  Luminal gain (MLD post-procedure - MLD pre-procedure)
In-stent MLD | 13 months - US patients only
  In-stent MLD
In-segment MLD | 13 months - US patients only
  In-segment (+5mm from the stent edges) MLD
In-segment late loss | 13 months - US patients only
  In-segment (+5mm from the stent edges) late loss
Proximal late loss | 13 months - US patients only
  Proximal late loss (+5 mm from proximal stent edge)
Distal late loss | 13 months - US patients only
  Distal late loss (+5 mm from proximal stent edge)
In-stent and in-segment Binary Restenosis | 13 months - US patients only
  In-stent and in-segment Binary Restenosis
OCT-determined inner layer percent neointimal hyperplasia volume | 13 months - US patients only
  OCT-determined inner layer percent neointimal hyperplasia volume
In-stent MLA | 13 months - US patients only
  In-stent MLA
In-segment minimum lumen area (MLA) | 13 months - US patients only
  In-segment minimum lumen area (MLA)
Minimal stent area (MSA) | 13 months - US patients only
  Minimal stent area (MSA)
Stent expansion | 13 months - US patients only
  Stent expansion
Edge dissection | 13 months - US patients only
  Edge dissection
% NIH at the MLA | 13 months - US patients only
  % NIH at the MLA
% Area stenosis at the MLA | 13 months - US patients only
  % Area stenosis at the MLA
Luminal gain (MLA post-procedure - MLA pre-procedure) | 13 months - US patients only
  Luminal gain (MLA post-procedure - MLA pre-procedure)
In-stent late loss MLA | 13 months - US patients only
  In-stent late loss MLA
In-segment (+5 mm from the stent edges) late loss (MLA). | 13 months - US patients only
  In-segment (+5 mm from the stent edges) late loss (MLA).
Proximal late loss (+5 mm from proximal stent edge) (MLA) | 13 months - US patients only
  Proximal late loss (+5 mm from proximal stent edge) (MLA)
Distal late loss (+5 mm from distal stent edge) (MLA) | 13 months - US patients only
  Distal late loss (+5 mm from distal stent edge) (MLA)
Intraluminal mass at least 0.2 mm beyond the luminal edge of a strut | 13 months - US patients only
  Intraluminal mass at least 0.2 mm beyond the luminal edge of a strut (Intraluminal mass attached to the vessel is defined as an irregularly shaped structure in contact with the luminal contour, a free intraluminal mass is defined as an isolated structure in the lumen without contact to the vessel wall)
Malapposition | 13 months - US patients only
  Malapposition (stent struts clearly separated from the vessel wall (lumen border/plaque surface) without tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm not associated with any side branch)
% Covered strut | 13 months - US patients only
  % Covered strut (NIH thickness of >0 μm).
% Healthy covered strut | 13 months - US patients only
  % Healthy covered strut (NIH thickness≥40 μm).
Peri-strut low intensity area | 13 months - US patients only
  Peri-strut low intensity area (peri-strut region of homogeneous lower intensity observed without signal attenuation).
Healing score | 13 months - US patients only
  Healing score (defined as % intraluminal mass [=intraluminal mass volume/stent volume] ×4 + % malposed and uncovered struts
  ×3 + (% uncovered struts alone ×2 + % malposed struts alone ×1) at 13 months.
  1. Intraluminal mass (+4).
  2. Malposed and uncovered struts (+3).
  3. Uncovered struts alone (+2).
  4. Malposed struts alone (+1).

CONTACTS AND LOCATIONS:
Locations (1):
- St Francis Hospital Heart Center, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No